CLINICAL TRIAL: NCT04617444
Title: Substudy of Efficacy, Safety and Toxicology of Electronic Nicotine Delivery Systems as an Aid for Smoking Cessation (ESTxENDS Trial)- the Olfactory Function Substudy of ESTxENDS
Brief Title: The ESTxENDS Trial- Substudy on Effects of Using Electronic Nicotine Delivery Systems (ENDS) on Olfactory Function
Acronym: ESTxENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Lausanne (Other); University of Geneva, Switzerland (Other); University of Zurich (Other); State Hospital, St. Gallen (Other Government); Swiss National Science Foundation (Other); Krebsforschung Schweiz, Bern, Switzerland (Other); Federal Office of Public Health, Switzerland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-02332j
Record Dates: First submitted 2020-10-24; First posted 2020-11-05 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation; Olfactory Disorder
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Masking Description: Statisticians and laboratory personnel will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: ENDS (vaporizer/e-cig) and smoking cessation counseling
- Control group (Active Comparator)
  Interventions: Other: Smoking cessation counseling

INTERVENTIONS:
Other: ENDS (vaporizer/e-cig) and smoking cessation counseling — Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Intervention group
Other: Smoking cessation counseling — Participants in the control group will receive smoking cessation counseling only. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Control group

SUMMARY:
--> This is a substudy of the main ESTxENDS trial (NCT03589989). Olfactory function outcomes should be considered secondary outcomes of the main smoking cessation outcome formulated in NCT03589989.

Up to one in five people have suffered loss or impairment of their sense of smell, limiting their available information about the environment, including possible hazards (e.g. gas or smoke). An impaired sense of smell is strongly associated with smoking, but its prevalence in smokers has yet to be established. Since only a few prospective cohort studies among smokers have compared change in olfactory function in smokers, it is not known how much or how fast smoking may impair olfactory function. Some studies describe improvement in olfactory function among quitters, supporting anecdotal evidence from ex-smokers who say they regained their sense of smell over time. As far as the investigators know, no randomized controlled trial has tested the effects of a smoking cessation intervention on olfactory function.

A reliable and validated olfactory function test is the Burghart Sniffin' Sticks 16-item Identification-test, which is quick and easy to administer. 16 familiar odours will be presented to the participants, each for 3-4 seconds. After each odour the participant is asked to select the correct answer from 4 possible answers.

With increasing popularity of e-cigarettes, their effect on the olfactory function also needs to be assessed. It is known, that e-cigarettes produce toxic compounds such as carbonyl and aldehydes, what could impair the sense of smell - especially if the liquid-level is too low or the temperature on the coil is too hot. This is the source of a phenomenon called "dry-hit", which is said to leave a burnt taste or smell to be recognized by users. However, it is unclear if e-cigarettes users with an olfactory dysfunction can adequately recognize a "dry-hit". Therefore, the goal is to investigate the effects of smoking cessation and use of ENDS on olfactory function and the recognition of a "dry-hit" from a test e-cigarette.

For the main ESTxENDS trial (NCT03589989), cigarette smokers motivated to quit smoking cigarettes will be included. Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants in the control group will receive smoking cessation counseling only. All participants will be followed over a 24-month period. The primary objective is to assess changes in olfactory function from baseline to 6 months post target quit date (TQD) in cigarette smokers randomized to the intervention group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Persons aged 18 or older
* Currently smoking 5 or more cigarettes a day for at least 12 months
* Willing to try to quit smoking within the next 3 months,
* Persons providing a valid phone number, a valid email address and/or a valid postal address.

Exclusion Criteria:

* Known hypersensitivity or allergy to contents of the e-liquid
* Participation in another study with investigational drug within the 30 days preceding the baseline visit and during the present study where interactions are to be expected
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the scheduled study intervention, i.e. within the first 6-months of the study
* Persons having used ENDS or tobacco heating systems regularly in the 3 months preceding the baseline visit
* Persons having used nicotine replacement therapy (NRT) or other medications with demonstrated efficacy as an aid for smoking cessation such as varenicline or bupropion within the 3 months preceding the baseline visit
* Persons who cannot attend the 6- month follow-up visit for any reason
* Cannot understand instructions delivered in person or by phone, or otherwise unable to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Assessment of olfactory function- Baseline | Baseline
  Assessment of olfactory function with the Burghart Sniffin' Sticks 16-item Identification-test. The highest possible score is 16; the cut-off for hyposmia is 11 and cut-off for anosmia is 8.
Assessment of olfactory function- follow-up | 6 months post quit date]
  Assessment of olfactory function with the Burghart Sniffin' Sticks 16-item Identification-test. The highest possible score is 16; the cut-off for hyposmia is 11 and cut-off for anosmia is 8.

SECONDARY OUTCOMES:
Assessment of change of olfactory function | change from baseline to 6 months post quit date
  Assessment of change of olfactory function with the Burghart Sniffin' Sticks 16-item Identification-test. The highest possible score is 16; the cut-off for hyposmia is 11 and cut-off for anosmia is 8.
Assessment of dry-hit recognition | 6 months post quit date
  Assessment of dry-hit recognition. Participants will be given 2 ENDS to have them assess the probability of a dry-hit. The participants will be asked to rate the probability of a dry-hit in both ENDS as follows:
  1. Definitely (3 points)
  2. Probably (2 points)
  3. Probably not (1 points)
  4. Definitely not (0 points) 2 or 3 points will be interpreted as correctly identifying the ENDS generating a dry-hit.

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, Prof.Dr.med, Study Director — Berner Institut für Hausarztmedizin (BIHAM)
Locations (5):
- Switzerland (5):
  - Unisanté, Centre universitaire de médecine générale et santé publique, Université de Lausanne, Lausanne, Canton of Vaud
  - University Clinic for General Internal Medicine, Bern University Hospital, Bern
  - Département de médecine interne, Hôpitaux universitaires de Genève, Geneva
  - Lungenzentrum, Klinik für Pneumologie und Schlafmedizin, Kantonsspital St. Gallen, Sankt Gallen
  - Epidemiology, Biostatistics and Prevention Institute (EBPI), University of Zurich, Zurich

REFERENCES:
- [Background] Whitcroft KL, Hummel T. Clinical Diagnosis and Current Management Strategies for Olfactory Dysfunction: A Review. JAMA Otolaryngol Head Neck Surg. 2019 Sep 1;145(9):846-853. doi: 10.1001/jamaoto.2019.1728. PMID 31318413
- [Background] Neuland C, Bitter T, Marschner H, Gudziol H, Guntinas-Lichius O. Health-related and specific olfaction-related quality of life in patients with chronic functional anosmia or severe hyposmia. Laryngoscope. 2011 Apr;121(4):867-72. doi: 10.1002/lary.21387. Epub 2011 Feb 4. PMID 21298638
- [Background] Doty RL, Kamath V. The influences of age on olfaction: a review. Front Psychol. 2014 Feb 7;5:20. doi: 10.3389/fpsyg.2014.00020. eCollection 2014. PMID 24570664
- [Background] Mullol J, Alobid I, Marino-Sanchez F, Quinto L, de Haro J, Bernal-Sprekelsen M, Valero A, Picado C, Marin C. Furthering the understanding of olfaction, prevalence of loss of smell and risk factors: a population-based survey (OLFACAT study). BMJ Open. 2012 Nov 6;2(6):e001256. doi: 10.1136/bmjopen-2012-001256. Print 2012. PMID 23135536
- [Background] Schubert CR, Cruickshanks KJ, Fischer ME, Huang GH, Klein BE, Klein R, Pankow JS, Nondahl DM. Olfactory impairment in an adult population: the Beaver Dam Offspring Study. Chem Senses. 2012 May;37(4):325-34. doi: 10.1093/chemse/bjr102. Epub 2011 Nov 1. PMID 22045704
- [Background] Jung HJ, Shin IS, Lee JE. Olfactory function in mild cognitive impairment and Alzheimer's disease: A meta-analysis. Laryngoscope. 2019 Feb;129(2):362-369. doi: 10.1002/lary.27399. Epub 2018 Nov 22. PMID 30565695
- [Background] Ajmani GS, Suh HH, Wroblewski KE, Pinto JM. Smoking and olfactory dysfunction: A systematic literature review and meta-analysis. Laryngoscope. 2017 Aug;127(8):1753-1761. doi: 10.1002/lary.26558. Epub 2017 May 31. PMID 28561327
- [Background] Frye RE, Schwartz BS, Doty RL. Dose-related effects of cigarette smoking on olfactory function. JAMA. 1990 Mar 2;263(9):1233-6. PMID 2304239
- [Background] Siegel JK, Wroblewski KE, McClintock MK, Pinto JM. Olfactory dysfunction persists after smoking cessation and signals increased cardiovascular risk. Int Forum Allergy Rhinol. 2019 Sep;9(9):977-985. doi: 10.1002/alr.22357. Epub 2019 Jul 31. PMID 31365791
- [Background] Vennemann MM, Hummel T, Berger K. The association between smoking and smell and taste impairment in the general population. J Neurol. 2008 Aug;255(8):1121-6. doi: 10.1007/s00415-008-0807-9. Epub 2008 Jul 28. PMID 18677645
- [Background] Dinc AS, Sengezer T, Cayonu M, Sahin MM. Smoking cessation improves olfactory functions. Laryngoscope. 2020 Feb;130(2):E35-E38. doi: 10.1002/lary.27992. Epub 2019 Apr 5. PMID 30953390
- [Background] Hummel T, Kobal G, Gudziol H, Mackay-Sim A. Normative data for the "Sniffin' Sticks" including tests of odor identification, odor discrimination, and olfactory thresholds: an upgrade based on a group of more than 3,000 subjects. Eur Arch Otorhinolaryngol. 2007 Mar;264(3):237-43. doi: 10.1007/s00405-006-0173-0. Epub 2006 Sep 23. PMID 17021776
- [Background] Rumeau C, Nguyen DT, Jankowski R. How to assess olfactory performance with the Sniffin' Sticks test((R)). Eur Ann Otorhinolaryngol Head Neck Dis. 2016 Jun;133(3):203-6. doi: 10.1016/j.anorl.2015.08.004. Epub 2015 Sep 4. PMID 26344139
- [Background] Farsalinos KE, Gillman G. Carbonyl Emissions in E-cigarette Aerosol: A Systematic Review and Methodological Considerations. Front Physiol. 2018 Jan 11;8:1119. doi: 10.3389/fphys.2017.01119. eCollection 2017. PMID 29375395
- [Background] Farsalinos KE, Voudris V, Poulas K. E-cigarettes generate high levels of aldehydes only in 'dry puff' conditions. Addiction. 2015 Aug;110(8):1352-6. doi: 10.1111/add.12942. Epub 2015 May 20. PMID 25996087
- [Derived] Walchli C, Grunig V, Tal K, Rodondi N, Berlin I, Humair JP, Frei A, Pohle S, Jakob J, Auer R, Poletti SC, Schoeni A. Association between duration or intensity of tobacco smoking and olfactory function: A cross-sectional study among smokers willing to quit smoking. Tob Induc Dis. 2025 Dec 20;23. doi: 10.18332/tid/211073. eCollection 2025. PMID 41424768